CLINICAL TRIAL: NCT06903949
Title: Comparison of the Analgesic Efficacy of Radiofrequency Application to Lumbar Root Ganglia in Geriatric and Young Patients With Chronic Radicular Lumbar Pain
Brief Title: Radiofrequency for Chronic Radicular Lumbar Pain: Geriatric vs. Young Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Turan, MD, Principal Investigator, Ankara Etlik City Hospital
Other Study IDs: Geriatric vs Young DRG
Record Dates: First submitted 2025-03-24; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Radiculopathy Lumbar; Radiculopathy, Lumbosacral Region; Chronic Pain
Keywords: Radiculopathy Lumbar; Radiculopathy, Lumbosacral Region; Chronic Pain
MeSH Terms: conditions — Radiculopathy; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young: Young group (18-64 years): These patients undergo Pulsed Radiofrequency therapy at the lumbar dorsal root ganglia, with treatment response and opioid consumption assessed post-procedure.
  Interventions: Procedure: Lumbar Dorsal Root Ganglia Pulsed Radiofrequency
- Geriatric: Geriatric group (≥65 years): These patients undergo Pulsed Radiofrequency therapy at the lumbar dorsal root ganglia, with treatment response and opioid consumption assessed post-procedure.
  Interventions: Procedure: Lumbar Dorsal Root Ganglia Pulsed Radiofrequency

INTERVENTIONS:
Procedure: Lumbar Dorsal Root Ganglia Pulsed Radiofrequency — It is an interventional pain management technique used to treat chronic radicular pain, often associated with conditions like lumbar disc herniation or degenerative disc disease. It involves the application of pulsed radiofrequency energy to the dorsal root ganglia (DRG), which are clusters of nerve cell bodies located just outside the spinal cord. DRG is involved in transmitting sensory signals from the periphery (e.g., the limbs) to the central nervous system.

SUMMARY:
This study aims to evaluate the treatment response and lumbar magnetic resonance imaging (MRI) findings of patients who have undergone pulsed radiofrequency therapy for chronic radicular lumbar pain at the dorsal root ganglia. By comparing young (18-64 years) and geriatric (≥65 years) patient groups, the study seeks to assess the impact of age on treatment response and opioid consumption. Additionally, it aims to analyze the potential relationship between paraspinal muscle fat infiltration and treatment outcomes.

DETAILED DESCRIPTION:
Chronic radicular lumbar pain is a significant health issue due to its increasing prevalence and impact on healthcare costs. Therefore, investigating and managing modifiable risk factors associated with chronic radicular lumbar pain play a crucial role in reducing the burden of this condition at both individual and societal levels. The most common causes of chronic radicular lumbar pain include intervertebral disc pathologies, facet joint degeneration, spinal canal stenosis, and mechanical or inflammatory involvement of neural structures. In cases resistant to medical and conservative treatment, interventional pain management techniques become the primary approach, making these patients the most frequently treated group in pain clinics.

Pulsed radiofrequency (PRF) therapy applied to the dorsal root ganglia (DRG) is a widely used minimally invasive interventional technique for radicular lumbar pain. In this procedure, fluoroscopy-guided insertion of specialized radiofrequency needles through the vertebral foramina allows the application of pulsed radiofrequency to the DRG. This technique modulates peripheral nociceptive signal transmission, contributing to pain relief.

Lumbar paraspinal muscles play a crucial role in maintaining spinal stability. Research on chronic low back pain suggests that fat infiltration in the paraspinal muscles is a significant factor in its pathophysiology. Lumbar magnetic resonance imaging (MRI) can be used to assess paraspinal muscle fat infiltration, which has been associated with higher pain intensity and poorer functional outcomes. The Goutallier classification is commonly used to grade fat infiltration. Previous studies suggest that in elderly patients with chronic low back pain, severe fat infiltration in the paraspinal muscles may be associated with a poor analgesic response to epidural steroid injections.

This study aims to evaluate the treatment response and lumbar MRI findings of patients who have undergone pulsed radiofrequency therapy for chronic radicular lumbar pain at the dorsal root ganglia. By comparing young (18-64 years) and geriatric (≥65 years) patient groups, the study seeks to assess the impact of age on treatment response and opioid consumption. Additionally, it aims to analyze the potential relationship between paraspinal muscle fat infiltration and treatment outcomes.

The medical records of patients who underwent pulsed radiofrequency therapy at the lumbar dorsal root ganglia will be reviewed retrospectively. Patients will be categorized into young (18-64 years) and geriatric (≥65 years) groups. Treatment efficacy will be assessed by retrospectively comparing Numeric Rating Scale (NRS) pain scores recorded before the procedure and at the 3rd month follow-up visit.

Since this is a retrospective study, the analysis will be conducted using existing clinical data without altering patient management or treatment plans. Additionally, pre-procedural lumbar MRI scans will be examined, and paraspinal muscle fat infiltration will be graded using the Goutallier classification. Demographic and clinical variables that may be associated with treatment response and paraspinal fat infiltration (including age, sex, body mass index (BMI), comorbidities, symptom duration, and opioid use) will be obtained from patient records.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older patients
* Patients that diagnosed with chronic radicular lumbar pain
* Have not received adequate response despite conservative treatments
* Have complete medical data available in the hospital data system

Exclusion Criteria:

* Missing data in the patient's follow-up records
* The patient has previously undergone interventional pain management
* The patient has previously had lumbar surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients who underwent pulsed radiofrequency (PRF) therapy at the lumbar dorsal root ganglia for chronic radicular lumbar pain. Participants are divided into two age groups: young group (18-64 years) and geriatric group (65 years and older). Only patients who have not responded well to medical and conservative treatments for their chronic radicular lumbar pain and have not undergone prior surgery will be included.
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale | Change from baseline to third month after treatment
  Numeric Rating Scale is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
Goutallier Classification | Pre-procedure grade
  The Goutallier grading system is a scale used to assess the degree of fat infiltration in the paraspinal muscles, typically evaluated through magnetic resonance imaging (MRI). Scores range from 0 (no fat infiltration, normal muscle) to 4 (complete fat infiltration, muscle entirely replaced by fat).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Ankara, Etlik, Turkey (Türkiye)